CLINICAL TRIAL: NCT03175952
Title: Virtual Histology Intravascular Ultrasound to Evaluate Prognostic Risks of Saphenous Vein Graft Disease Before Percutaneous Coronary Intervention.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Chest Hospital (Other)
Responsible Party: Principal Investigator, Yin Liu, director, Cardiology Department, Tianjin Chest Hospital
Other Study IDs: 16YFZCSY00800
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Major Adverse Cardiovascular Events; Saphenous Vein Graft Disease; Virtual Histology Intravascular Ultrasound; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCI
  Interventions: Diagnostic Test: virtual histology intravascular ultrasound

INTERVENTIONS:
Diagnostic Test: virtual histology intravascular ultrasound — Patients with saphenous vein graft disease will be examined using virtual histology intravascular ultrasound, and treated with percutaneous coronary intervention. Then they will be followed up at 1, 6 and 12 months.
  Other Names: percutaneous coronary intervention

SUMMARY:
The study is a prospective cohort study conducted in Tianjin Chest Hospital, China. Patients with saphenous vein graft disease after coronary artery bypass graft, and planning for receiving percutaneous coronary intervention after virtual histology intravascular ultrasound will be enrolled between May 2017 and April 2019. These subjects will be followed up at 1, 6 and 12 months post-operation of PCI to assess the short-term and long-term effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SVGD after CABG
* Planning to receive PCI using drug-eluting stents
* 18 to 80 years old
* Finishing VH-IVUS examination
* Willing to participate in the study and sign informed consent

Exclusion Criteria:

* Patients with liver disfunction and renal failure
* Aspirin and clopidogrel allergy
* Acute myocardial infarction after CABG
* History of stroke in the past 3 months
* Gastrointestinal bleeding and hemoptysis recently
* Vasculitis and non-atherosclerotic coronary artery disease
* Coagulation disorders
* History of malignancy
* Women during pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is a prospective cohort study conducted in Tianjin Chest Hospital, China. Patients with SVGD after CABG, and planning for receiving PCI after VH-IVUS will be enrolled between April 2017 and March 2019. These subjects will be followed up at 1, 6 and 12 months post-operation of PCI to assess the short-term and long-term effect.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular events | after PCI for saphenous vein graft disease (SVGD) in one year
  Cardiac death, myocardial infarction, target lesion revascularization and target vessel revascularization are all major adverse cardiovascular events

SECONDARY OUTCOMES:
Thrombolysis In Myocardial Infarction (TIMI) flow in 24 hours after PCI for the SVGD | 24 hours after PCI for the SVGD
Number of slow reflow, no reflow or distal embolization of the saphenous vein graft after PCI on the basis of Corrected TIMI Frame Count (TFC) | 24 hours after PCI for the SVGD
Success rate of PCI | 24 hours after PCI for the SVGD
  The residual stenosis of SVG is less than 50% and achieving TIMI flow 3

CONTACTS AND LOCATIONS:
Overall Officials: Yin Liu, Principal Investigator — Tianjin Chest Hospital
Locations (1):
- Tianjin Chest Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu Y, Wang HB, Li X, Xiao JY, Wang JX, Reilly KH, Sun B, Gao J. Relationship between plaque composition by virtual histology intravascular ultrasound and clinical outcomes after percutaneous coronary intervention in saphenous vein graft disease patients: study protocol of a prospective cohort study. BMC Cardiovasc Disord. 2018 Dec 12;18(1):233. doi: 10.1186/s12872-018-0975-1. PMID 30541457